CLINICAL TRIAL: NCT05100407
Title: Evaluation of the Prevalence and Antibiotic Susceptibility Pattern of Multidrug Resistance Bacteria and Its Association With Patients' Predictive Factors
Brief Title: Factors Impacting the Prevalence of MDR Bacteria
Status: Completed | Type: Observational
Sponsor: Kufa University (Other)
Responsible Party: Principal Investigator, Zahraa Najah Mohsin, general pharmacist, Kufa University
Other Study IDs: MDR and predictive factors
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-03

CONDITIONS: Multi-antibiotic Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To determine the prevalence of multidrug resistance bacteria in patient with different infections
2. To evaluate patients' predictive risk factors of antimicrobial resistance
3. To assess the association between patients' factors and prevalence of MDR bacteria

DETAILED DESCRIPTION:
Antimicrobial resistance is one of the most critical public health issue in this century . WHO declared antimicrobial resistance as one of the top ten global health threats that impend the effective management and prevention of evolving infections .

Antimicrobial resistance nowadays poses a big challenge because of the emerging of resistance to the antibiotics that previously effective and development of multidrug resistance infections with subsequent increase in morbidity, mortality and financial loss .

In spite of WHO health strategies that taken to face multidrug resistance problem, the burden of antimicrobial resistance in Europe is compared with combined burden of influenza and HIVS .while in USA the estimated antibiotics resistance infections is 2.8 millions and the related deaths exceeded 35,000 every year and expected to reach to ten million deaths with collective cost of 100 trillion USD annually in 2050 .

Numerous studies reported that self-medications, improper prescription, overuse of antibiotics, deficiency of antibiotics susceptibility test and limited knowledge and attitude of population towards antibiotics are the main factors that lead to antibiotics efficacy being reduced with long hospital stay. Other studies stated that the predictive indicators of MDR tragedy are age, gender, comorbidities, previous hospital stay or antibiotic use .

In low and middle income countries like IRAQ there is a difficulty in estimation the scope of antibiotics resistance problem and its evolving over time due to the lack of surveillance, besides alarmingly excessive antibiotics consumption added other challenges and urged us to aim this study .

ELIGIBILITY:
Inclusion Criteria:

* patients who were screened for MDR bacteria
* patients who accepted to participate in the study

Exclusion Criteria:

* patients with no growth media
* patients who cannot communicated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients hospitalized with bacterial infection and screened for MDR bacteria in AL-Zahraa teaching hospital or AL-Sader medical city
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of multidrug resistance bacteria in isolated patient specimen | based line value (zero months)
  proportion of MDR bacteria that detected in isolated specimen
Association of patient's factors with prevalence of multidrug resistance Bacteria. | based line value (zero months)
  exploring the association between patient's factors and the prevalence of MDR bacteria by multivariate analysis

SECONDARY OUTCOMES:
Prevalence of Methicillin resistance staph. Aureus (MERSA) | based line value (zero months)
  proportion of participants with MERSA bacteria that detected in isolated specimen
Prevalence of vancomycin (-resistant Enterococci VRE) | based line value (zero months)
  proportion of participants with VRE bacteria that detected in isolated specimen
Prevalence of extended spectrum β lactamase producers (ESBL) | based line value (zero months)
  proportion of participants with ESBL bacteria that detected in isolated specimen
Knowledge, attitude and practice (KAP) toward antibiotic use | based line value (zero months)
  the score indicator of KAP through a module of KAP survey by 20 categorized questions the knowledge is individual understanding about antibiotic resistance the attitude is the perceptions and beliefs that respondents (+),(-) perceive towards antibiotic resistance the practice is the observable actions of individual towards antibiotic use
Risk factors for antibiotic resistance | based line value (zero months)
  asses patient's predictive factors and their role in prevalence of multidrug resistance bacteria

CONTACTS AND LOCATIONS:
Overall Officials: Hayder Asaad, assist. prof, Study Director — college of pharmacy kufa university
Locations (1):
- Faculty of pharmacy /kufa university, Najaf, Iraq

REFERENCES:
- [Background] Prestinaci F, Pezzotti P, Pantosti A. Antimicrobial resistance: a global multifaceted phenomenon. Pathog Glob Health. 2015;109(7):309-18. doi: 10.1179/2047773215Y.0000000030. Epub 2015 Sep 7. PMID 26343252
- [Background] Who.int. 2021. Antimicrobial resistance. [online] Available at: https://www.who.int/health-topics/antimicrobial-resistance
- [Background] Bhardwaj, K., Shenoy M, S., Baliga, S., Unnikrishnan, B. and Baliga, B., 2021. Knowledge, attitude, and practices related to antibiotic use and resistance among the general public of coastal south Karnataka, India - A cross-sectional survey. Clinical Epidemiology and Global Health, 11, p.100717
- [Background] Mallah N, Rodriguez-Cano R, Figueiras A, Takkouche B. Design, reliability and construct validity of a Knowledge, Attitude and Practice questionnaire on personal use of antibiotics in Spain. Sci Rep. 2020 Nov 26;10(1):20668. doi: 10.1038/s41598-020-77769-6. PMID 33244041
- [Background] Marzan M, Islam DZ, Lugova H, Krishnapillai A, Haque M, Islam S. Knowledge, Attitudes, and Practices of Antimicrobial Uses and Resistance Among Public University Students in Bangladesh. Infect Drug Resist. 2021 Feb 11;14:519-533. doi: 10.2147/IDR.S289964. eCollection 2021. PMID 33603416
- [Background] Rodriguez-Villodres A, Martin-Gandul C, Penalva G, Guisado-Gil AB, Crespo-Rivas JC, Pachon-Ibanez ME, Lepe JA, Cisneros JM. Prevalence and Risk Factors for Multidrug-Resistant Organisms Colonization in Long-Term Care Facilities Around the World: A Review. Antibiotics (Basel). 2021 Jun 7;10(6):680. doi: 10.3390/antibiotics10060680. PMID 34200238
- [Background] Lim C, Takahashi E, Hongsuwan M, Wuthiekanun V, Thamlikitkul V, Hinjoy S, Day NP, Peacock SJ, Limmathurotsakul D. Epidemiology and burden of multidrug-resistant bacterial infection in a developing country. Elife. 2016 Sep 6;5:e18082. doi: 10.7554/eLife.18082. PMID 27599374